CLINICAL TRIAL: NCT04195984
Title: Evaluation of the Efficacy and Safety of the Mi-thos® Transcatheter Mitral Valve Replacement System in Patients with Severe Mitral Valve Disease At High Surgical Risk.
Brief Title: Mi-thos® Transcatheter Mitral Valve Replacement Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai NewMed Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-valve-2018-06
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Mitral Valve Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Transcatheter mitral valve replacement with the Mi-thos® valve and transcatheter delivery system
  Interventions: Device: Mi-thos® valve and transapical delivery system

INTERVENTIONS:
Device: Mi-thos® valve and transapical delivery system — Transcatheter mitral valve replacement system

SUMMARY:
To evaluate the safety and performance of the Mi-thos® Mitral Heart Valve with the Mi-thos® Transcatheter Delivery System.

DETAILED DESCRIPTION:
The Mi-thos® study is an multicenter, single-arm, prospective, safety and performance clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Severe mitral valve regurgitation ≥ 3+;
* High surgical risk fot open mitral valve surgery;
* Age ≥ 65 years old;
* Life expectancy > 12 months;
* As assessed by multidisciplinary cardiac team, patients who are not eligible for surgery;
* Patients sign an informed consent form.

Exclusion Criteria:

* Previous cardiac mitral valve surgery;
* Active infections requiring antibiotic therapy;
* Clinically significant untreated Coronary Artery Disease (CAD);
* Pulmonary hypertension （Pulmonary systolic pressure > 70 mmHg）;
* Patients with severe right heart failure;
* Left ventricular ejection fraction <25%;
* Diagnosis of hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis;
* Dialysis patient;
* Patients with severe coagulopathy;
* Patients with contraindications to anticoagulant drugs;
* Patients with stroke or transient ischemic within 30 days;
* Echocardiography found any intracardiac mass, left ventricle or atrial thrombus;
* Patients who require surgery or interventional therapy for other valvular lesions;
* Patients with severe macrovascular disease requiring surgical treatment;
* Patients with more than 70% of carotid stenosis;
* To be allergic to contrast agents, nickel-titanium memory alloys or bovine-derived products;
* Patients with severe neurological disorders affecting cognitive ability;
* Patients with severe thoracic deformities.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from all-cause mortality | 1 year
  All-cause mortality after TMVR

SECONDARY OUTCOMES:
Freedom from all-cause mortality | 30 days, 6months, 2-5 years
  All-cause mortality after TMVR
Severe adverse event rate | 30 days, 6months, 1 year, 2-5 years
  Severe adverse events rate after TMVR
NYHA Heart Function Rating | 30 days, 6months, 1 year, 2-5 years
  NYHA Heart Function Rating after TMVR
Kansas City Cardiomyopathy score | 30 days, 6months, 1 year, 2-5 years
  Kansas City Cardiomyopathy score after TMVR

CONTACTS AND LOCATIONS:
Overall Officials: Wang chunsheng, Chief, Principal Investigator — Shanghai Zhongshan Hospital
Locations (3):
- China (3):
  - Fuwai hospital, Beijing, Beijing Municipality
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Xijing hospital, Xi’an, Shanxi